CLINICAL TRIAL: NCT00591617
Title: Optimizing Outcomes Using Suboxone for Opiate Dependence
Acronym: OpBup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Walter Ling, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA020210 (NIH)
Record Dates: First submitted 2007-12-28; First posted 2008-01-11 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Opioid Dependency
Keywords: Opioids; drug dependence; drug abuse; treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1: MM (Active Comparator): Medical Management: group receives medical management from study physician and Suboxone pharmacotherapy
  Interventions: Other: Psychosocial treatment plus Suboxone pharmacotherapy
- 2: CBT (Active Comparator): Cognitive Behavioral Therapy (CBT) group receives CBT, medical management and Suboxone pharmacotherapy
  Interventions: Other: Psychosocial treatment plus Suboxone pharmacotherapy
- 3: CM (Active Comparator): Contingency Management (CM) group receives CM, medical management, and Suboxone pharmacotherapy
  Interventions: Other: Psychosocial treatment plus Suboxone pharmacotherapy
- 4: CBT + CM (Active Comparator): Cognitive Behavioral Therapy (CBT) and Contingency Management (CM) group receives CBT, CM, medical management, and Suboxone pharmacotherapy
  Interventions: Other: Psychosocial treatment plus Suboxone pharmacotherapy

INTERVENTIONS:
Other: Psychosocial treatment plus Suboxone pharmacotherapy — Participants randomly assigned to one of four psychosocial treatment conditions building on pharmacotherapy with Suboxone (buprenorphine + naloxone)

SUMMARY:
Building on a platform of pharmacological treatment with Suboxone (buprenorphine and naloxone), participants are randomly assigned to one of four psychosocial treatment conditions.

DETAILED DESCRIPTION:
The approval of buprenorphine (combined with naloxone as Suboxone®) by the FDA enables physicians in the United States to provide pharmacotherapy treatment to opioid-dependent patients in private medical settings. Buprenorphine's wide acceptance and implementation by physicians has been slower than expected, however, and this may be due in part to the nature and necessity of providing comprehensive treatment for opioid-dependent patients. Lessons learned from methadone maintenance make it clear that simply providing opioid substitution does not address the behavioral components of dependence. While there is no lack of behavioral treatment facilities for substance abuse in the United States, what is lacking is an integrative approach to the treatment of opioid dependence using pharmacotherapy in conjunction with proven behavioral treatment strategies. Following a two-week stabilization and baseline period, this project will randomize 240 participants into 4 behavioral treatment groups featuring cognitive behavioral therapy and contingency management therapy. A universal, manual-guided psychosocial standard of care for buprenorphine pharmacological treatment allows for ethical inclusion of a "no-CBT or CM therapy" condition and closely resembles the current standard of psychosocial care delivered with opioid treatment using Suboxone®. Behavioral therapies will be delivered for 16 weeks (to study week 18) in conjunction with continued care with Suboxone®. An additional 16 weeks of treatment using Suboxone® (to study week 34) will ensue during which no CBT or CM therapies are provided. All participants enter a buprenorphine taper and return at study week 52 for long-term follow-up evaluations. Outcomes for the trial include illicit drug use (urine drug samples collected three times per week during the first 18 weeks), drug craving, retention (days in the protocol), psychiatric status (depression, mood), HIV risk behaviors, and treatment feasibility ratings. Results will be used to recommend strategies to optimize buprenorphine treatment outcomes and promote integration of pharmacotherapy and psychosocial/behavioral treatment strategies for physicians and for behavioral treatment facilities treating opioid-dependent patients.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Be 15 years of age or older.
2. Meet DSM-IV-TR criteria for opioid dependence.
3. Be interested in receiving buprenorphine treatment for their opioid dependence.
4. Be in good general health or, in case of a medical/psychiatric condition needing ongoing treatment, be under the care of a physician who provides documented willingness to continue participant's medical management and coordinate care with the study physicians. *
5. Be agreeable to and capable of signing an informed consent.
6. Have means of reliable transportation over the study period.
7. If female and of child bearing potential, agree to use of one of the following methods of birth control or be surgically sterile:

   1. oral contraceptives
   2. patch
   3. barrier (diaphragm or condom)
   4. intrauterine contraceptive system
   5. levonorgestrel implant
   6. medroxyprogesterone acetate contraceptive injection
   7. complete abstinence from sexual intercourse
   8. hormonal vaginal contraceptive ring
8. Be agreeable to and capable of complying with study procedures.

Exclusion Criteria:

Participants must not:

1. Have a known sensitivity to buprenorphine or naloxone.
2. Be dependent on alcohol, benzodiazepines or other drugs of abuse that require immediate medical attention.
3. Have a medical condition that would, in the opinion of the study physician, make participation medically hazardous (e.g., acute hepatitis, unstable cardiovascular, liver or renal disease).
4. Have a current pattern of benzodiazepine use, as assessed by the study physician, which would preclude safe participation in the study.
5. Be actively involved in another clinical trial.
6. Be acutely psychotic, severely depressed, and in need of inpatient treatment, or is an immediate suicide risk.
7. Be a nursing or pregnant female. Females who become pregnant during the course of the study will be withdrawn from the study and referred to an appropriate treatment venue; i.e. narcotic treatment program or specialty addiction clinic.
8. Be a female of childbearing potential who does not agree to use a medically acceptable method of birth control, e.g. oral contraceptives, barrier (diaphragm or condom) with or without spermicide, levonorgestrel implant, intra-uterine progesterone contraceptives system, medroxyprogesterone acetate contraceptive injection, or complete abstinence.
9. Have any pending legal action that could prohibit continued participation for the one-year period of study participation (such as that which could possibly result in incarceration).
10. Be expecting to leave the clinic's geographic area prior to study completion (within one year).
11. Have been previously randomized to a treatment condition in this study. -

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2006-09; Primary Completion 2012-01 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Comparison the effectiveness of four psychosocial treatment conditions as measured by self-reported abstinence from opioids verified by urine toxicology tests | Week 18 - At end of first phase

SECONDARY OUTCOMES:
Comparison across treatment conditions for reducing the severity of opioid-related problems | at end of Phase 1 (wk 18), phase 2 (wk 34) and two follow-up timepoints (wks. 40 and 52)
Comparison across treatment conditions for reducing the proportion of use-days of other substances of abuse (alcohol, marijuana, amphetamines, methamphetamines, benzodiazepines and barbiturates) as determined by self-report and urine test results. | At end of Phase 1 (wk. 18), Phase 2 (wk. 34), and at two follow-ups (wks. 40 and 52)
Comparison across treatment conditions in reducing psychiatric and mood disturbance as measured with the BDI and SF-36. | At end of Phase 1 (wk. 18), Phase 2 (wk. 34), and at two follow-ups (wks. 40 and 52)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — UCLA Integrated Substance Abuse Programs; Maureen Hillhouse, Ph.D., Study Director — UCLA Integrated Substance Abuse Programs
Locations (1):
- UCLA Integrated Substance Abuse Programs Outpatient Clinical Research Center, Los Angeles, California, United States

REFERENCES:
- [Derived] McHugh RK, Bailey AJ, McConaghy BA, Weiss RD, Fiellin DA, Hillhouse M, Moore BA, Fitzmaurice GM. Behavioral Therapy as an Adjunct to Buprenorphine Treatment for Opioid Use Disorder: A Secondary Analysis of 4 Randomized Clinical Trials. JAMA Netw Open. 2025 Aug 1;8(8):e2528529. doi: 10.1001/jamanetworkopen.2025.28529. PMID 40833692
- [Derived] Nielsen S, Hillhouse M, Mooney L, Fahey J, Ling W. Comparing buprenorphine induction experience with heroin and prescription opioid users. J Subst Abuse Treat. 2012 Oct;43(3):285-90. doi: 10.1016/j.jsat.2011.12.009. Epub 2012 Feb 1. PMID 22301084